CLINICAL TRIAL: NCT06747117
Title: STRIDE II: A Study of Patients With Lower Extremity Acute Limb Ischemia to Remove Thrombus With the Indigo™ Aspiration System II
Brief Title: A Study of Patients With Lower Extremity Acute Limb Ischemia to Remove Thrombus With the Indigo™ Aspiration System (STRIDE II)
Acronym: STRIDE II
Status: Recruiting | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 30000
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lower Extremity Acute Limb Ischemia; LE ALI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with lower extremity acute limb ischemia: Device: Indigo Aspiration System
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — Mechanical aspiration thrombectomy with the Indigo Aspiration System.

SUMMARY:
The primary objective of this study is to collect and evaluate clinical evidence supporting the safety and performance of the Indigo™ Aspiration System in a patient population with lower extremity acute limb ischemia (LE ALI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with a confirmed diagnosis of lower limb arterial occlusion located in the common iliac or below, with a minimum of 2 cm of proximal patency in the common iliac
* Acute occlusion with symptom duration of 14 days or less at presentation
* ALI Rutherford Category I, IIa or IIb
* First-line treatment with the Indigo Aspiration System using Computer Assisted Vacuum Thrombectomy (CAVT) aspiration tubing
* Informed consent is obtained from either patient or legally authorized representative (LAR) per Institutional Review Board/Ethics Committee requirements
* Previously enrolled patients presenting with a new acute occlusion in the contralateral limb meeting all eligibility criteria may be re-enrolled if the new acute occlusion is greater than 30 days from the initial index procedure

Exclusion Criteria:

* Life expectancy <1 year
* Target vessel size <2 mm
* Target thrombus is in the aorta or isolated profunda artery
* Prior major amputation (proximal to the tarsometatarsal joint) in the target limb
* Prior minor amputation in the target limb within the past 6 months that is not completely healed or cannot bear weight
* LE ALI secondary to dissection, vasculitis, or target vessel trauma, including iatrogenic etiology from treatment of a proximal location in the target limb
* Target thrombus in a saphenous vein bypass graft
* Treatment of the index event with thrombolytics or any other endovascular or open surgical method prior to enrollment
* Pregnancy
* Contraindication or sensitivity to iodinated intravascular contrast that cannot be adequately premedicated
* Other medical, behavioral, or psychological conditions that, in the opinion of the Investigator, precludes the patient from appropriate consent, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
* Current participation in another investigational drug or device study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present with LE ALI who are eligible for mechanical thrombectomy using the Indigo Aspiration System
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Target Limb Salvage Rate | 30 Days Post-Procedure

SECONDARY OUTCOMES:
Technical Success | Immediate Post Procedure
  Technical success defined as Thromboaspiration in Peripheral Ischemia (TIPI) 2/3 flow immediately post procedure by physician visual assessment of intraprocedural angiography
Primary Patency at 30 Days | 30 Days Post-Procedure
Rates of Device-related Major Bleeding | Procedure, 30 Days, and 180 Days Post-Procedure
Rates of Device-related Distal Embolization | During Procedure
Rates of Device-related Serious Adverse Events (SAE) | Procedure, 30 Days, and 180 Days Post-Procedure
Mortality | 30 Days and 180 Days Post-Procedure
  All cause mortality at 30 and 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — Vanderbilt University Medical Center; Dierk Scheinert, MD, Principal Investigator — Universitätsklinik Leipzig
Locations (23):
- United States (19):
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Community Memorial Hospital, Ventura, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Baptist Hospital of Miami, Miami Cardiac and Vascular Institute, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Community Hospital, Munster, Indiana
  - University of Maryland, Baltimore, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Health, New York, New York
  - TriHealth Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Flinders Medical Centre, Bedford Park, South Australia, Australia
- Universitätsklinik Leipzig, Leipzig, Germany
- ASST Degli Spedali Civili di Brescia, Brescia, Italy
- Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No